CLINICAL TRIAL: NCT03639558
Title: TREC-Lebanon Trial: A Randomised Controlled Trial for Rapid Tranquilisation for Agitated Patients in the Emergency Setting
Brief Title: TREC-Lebanon: A Trial for Rapid Tranquilisation for Agitated Patients in the Emergency Setting
Acronym: TREC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joseph Dib (Other Government)
Collaborators: University of Nottingham (Other); Hopital Psychiatrique De La Croix (Other Government)
Responsible Party: Sponsor-Investigator, Joseph Dib, Director of Trial Research, Hopital Psychiatrique De La Croix
Organization: Hopital Psychiatrique De La Croix (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPAP - 2018 - 0138 - 1
Record Dates: First submitted 2018-08-15; First posted 2018-08-21 (Actual); Results first posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Psychiatric Emergency; Aggression; Agitation
MeSH Terms: conditions — Aggression; Psychomotor Agitation | interventions — Haloperidol; Promethazine; Chlorpromazine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Haloperidol + Promethazine + Chlorpromazine (Active Comparator): Haloperidol + Promethazine + Chlorpromazine are all psychiatric drugs that have been well tested. The combination of these 3 drugs, however, have never been randomised.
  Interventions: Drug: Haloperidol + Promethazine + Chlorpromazine
- Haloperidol + Promethazine (Experimental): Haloperidol + Promethazine are both psychiatric drugs with antipsychotic and calming properties.
  Interventions: Drug: Haloperidol + Promethazine

INTERVENTIONS:
Drug: Haloperidol + Promethazine + Chlorpromazine — This is the usual treatment given by this hospital during an aggressive psychiatric episode.
  Other Names: HPC
  Arms: Haloperidol + Promethazine + Chlorpromazine
Drug: Haloperidol + Promethazine — This is the second most used psycho-pharmacological combination used in this hospital during an aggressive psychiatric episode.
  Other Names: HP
  Arms: Haloperidol + Promethazine

SUMMARY:
This is a randomised controlled trial comparing haloperidol + promethazine versus haloperidol + promethazine + chlorpromazine for agitated patients in the emergency department.

DETAILED DESCRIPTION:
This is a randomised controlled trial comparing haloperidol + promethazine versus haloperidol + promethazine + chlorpromazine for agitated patients in the emergency department. Around 10% of patients will present to the psychiatric emergency unit with a violent episode that requires rapid tranquilisation. Surveys of practice and opinion has shown that variety of methods have been used and no universal option exists. This study will look at Haloperidol plus promethazine versus haloperidol plus promethazine plus chlorpromazine in violent aggressive psychiatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be eligible if (1) requiring emergency acute intramuscular sedation because of disturbed and dangerous behaviour and (2) if the clinician is uncertain of the benefits between haloperidol plus promethazine vs haloperidol plus promethazine plus chlorpromazine.
* Gender - both male and female
* Age (18-64)
* Clinician is unaware on the effects of either treatment interventions

Exclusion Criteria:

* If the clinician KNOWS one treatment has benefit over another for a particular person
* If the clinician is aware of a contra-indication of one of the treatments
* If there is an Advanced Directive expressing a wish for one or other, or another treatment in the emergency setting.
* If the clinician does not want to undertake for both personal and professional reasons.
* If the participant is known to be allergic to one or more of the interventions
* Already randomized
* Already sedated
* Accompanying person (Friend/Family/Police Officer) refuses patient trial entry

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Lebanon (2):
  - Hôpital Psychiatrique De La Croix, Beirut, Jal L Dib
  - Psychiatric Hospital of the Cross, Beirut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dib JE, Adams CE, Ikdais WH, Atallah E, Yaacoub HE, Merheb TJ, Kazour F, Tahan F, Haddad G, Zoghbi M, Azar J, Haddad C, Hallit S. Study protocol for a randomised controlled trial of haloperidol plus promethazine plus chlorpromazine versus haloperidol plus promethazine for rapid tranquilisation for agitated psychiatric patients in the emergency setting (TREC-Lebanon). F1000Res. 2019 Aug 15;8:1442. doi: 10.12688/f1000research.19933.1. eCollection 2019. PMID 32528650

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
Started | 52 | 48
Completed | 51 | 43
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 52 | 48 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of participant
  Years | 37 (11.4) | 36 (12.3) | 36 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 5 withdrawn from follow up citing unwillingness to be involved in the trial.
  1 withdrawn from hospital care by relevant authorities.
  Participants
    number analyzed (Participants) | 51 | 43 | 94
    Female | 27 | 22 | 49
    Male | 24 | 21 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 52 | 48 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to the Time Taken for Aggressive Behaviour to Change to Calm and Tranquil
Description: Patient no longer exhibiting aggressive behavior both verbal and physical post intervention treatment. A primary measure of outcome form will contain a Calm or Tranquil column followed by four rows: 20 mins, 40 mins, 60 mins and 120 mins post intervention medication. The boxes would be ticked depending if the patient meets the primary measure of outcome within the time frame provided.
Time Frame: 20, 40, 60 and 120 minutes post intervention treatment
Measure: Number; unit: participants
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
Number analyzed (Participants) | 52 | 48
participants
  Calm or tranquil at 20 minutes | 18 | 14
  Calm or tranquil at 40 minutes | 41 | 25
  Calm or tranquil at 60 minutes | 45 | 35
  Calm or tranquil at 120 minutes | 47 | 35

2. Secondary Outcome: Time Taken for Patient to Fall Asleep Post Intervention
Description: Patient has fallen asleep and is no longer aggressive post intervention treatment and will be noted on the outcomes form which includes a checklist of different time intervals: 20, 40, 60 and 120 minutes post intervention treatment.
Time Frame: 20, 40, 60 and 120 minutes post intervention treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
Number analyzed (Participants) | 52 | 48
Participants
  Asleep at 20 minutes | 0 | 2
  Asleep at 40 minutes | 9 | 9
  Asleep at 60 minutes | 25 | 10
  Asleep at 120 minutes | 24 | 18

3. Secondary Outcome: Time Patient Was Placed in Straitjacket/Restraint Post Intervention Treatment
Description: If patient was placed in a straitjacket post intervention due to aggression - this would be noted on the outcomes form which includes a checklist at certain time intervals 20,40,60 and 120 minutes post intervention treatment.
Time Frame: 20, 40, 60 and 120 minutes post intervention treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
Number analyzed (Participants) | 52 | 48
Participants
  Restraints at 20 minutes | 17 | 16
  Restraints at 40 minutes | 10 | 13
  Restraints at 60 minutes | 8 | 9
  Restraints at 120 minutes | 6 | 5

4. Secondary Outcome: Time Noted Where Important Adverse Effects Occurred Post Intervention
Description: If patient exhibits any adverse effects post intervention treatment, this will be noted within the time frames.
Time Frame: 20, 40, 60 and 120 minutes post intervention treatment
Population: Total number of participants who were analysed for adverse effects post intervention. No patients exhibited adverse effects in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
Number analyzed (Participants) | 52 | 48
Participants | 0 | 0

5. Secondary Outcome: Time Patient Left the Ward Against Medical Advice During the Time Period After the Intervention Was Administered.
Description: If patient had to leave ward against medical advice during intervention phase - the time will be noted as well as the reason to why patient left.
Time Frame: 20, 40, 60 and 120 minutes post intervention treatment
Population: Data not collected.
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 10 months from time of intervention.
Description: No change of definitions pertaining to adverse events. No further relevant information to be provided.
Arm/Group | Haloperidol + Promethazine + Chlorpromazine | Haloperidol + Promethazine
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/48
Other Adverse Events (participants affected / at risk) | 0/52 | 0/48

LIMITATIONS AND CAVEATS:
Possible limitations for this trial are that there are no Emergency Departments; therefore residents must always carry the TREC envelopes at all times, increasing the risk for error (i.e. misplacing envelope, using wrong envelope, etc.). Despite the limitation, the chances of error remain low due to the small sample size of 100.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/58/NCT03639558/Prot_SAP_ICF_003.pdf